CLINICAL TRIAL: NCT05072353
Title: Autologous Adipose Tissue Harvested With Superficial Enhanced Fluid Fat Injection (SEFFICARE) Method for Treatment of Diabetic Foot Ulcer Undergoing Minor Amputation (SEFFIDiFA): Proposal of Basic Research and Prospective Observational Study
Brief Title: Effectiveness of the Autologous Adipose Tissue Harvested With SEFFICARE Method for Treatment of DFU Minor Amputation
Acronym: SEFFIDiFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Nicola Leone, MD, Azienda Ospedaliero-Universitaria di Modena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEFFIDiFA_vers1.0
Record Dates: First submitted 2021-09-10; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer; Amputation
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): DFU Patients are subjected to digital or transmetatarsal amputation. The treatment is provided during the amputation surgical session according to the SEFFI technique. The SEFFICARE® system (SEFFILINE S.r.l., Via delle Lame, 98, 40122 Bologna, Italy) is a disposable commercially available device. The device is provided in a sterile bag without any drugs. The SEFFI is a 5-step technique meaning preparation, anesthesia, harvesting, washing, and fluidification. The resulting tissue (2.5 mL per syringe) is ready for grafting. The stumps are closed by primary intention following adipose tissue injection.
  Interventions: Device: SEFFICARE

INTERVENTIONS:
Device: SEFFICARE — The SEFFI is a 5-step technique:
  1. Preparation: the lower/lateral abdomen is chosen as the donor site.
  2. Anesthesia: the donor site is injected with a local anesthetic.
  3. Harvesting: a 0.8 mm or 0.5 mm cannula connected to a 10-ml VacLok® syringe is used to harvest the adipose tissue. The total amount of the harvested tissue could vary from 10 to 30 mL.
  4. Washing: The syringe containing the lipoaspirate tissue is immediately filled with sterile physiological solution. After some minutes the syringes in the decanting stand will show a separation by the gravity of the tissue (top) from the physiological solution (bottom).
  5. Fluidification: the syringe containing the adipose tissue should be connected to an empty 10 ml syringe. After pushing the tissue about 3 times from one syringe to the other, a good fluidification of the tissue is obtained.
  The resulting tissue (2.5 mL per syringe) is ready for grafting the amputation wound.

SUMMARY:
Diabetic foot ulcers (DFU) are one of the complications of diabetes mellitus resulting from multiple causes such as neuropathy, ischemia, and infection that contribute to morbidity and amputation. The prevalence of DFU has been estimated to be 3 to 5 times higher than the overall population. Minor amputations (digital or transmetatarsal) are the treatment of choice in case of irreversible DFU. However, many minor amputations do not heal and require re-amputation. Improvements of healing rate after adipose stem cells (ASCs) injection through micro-fragmented autologous adipose tissue of the amputation stump following minor DFU amputation were demonstrated. The use of ASCs obtained from the superficial enhanced fluid fat injection technique (SEFFICARE) to improve the healing process after DFUs minor amputation is the object of the present study.

A single-center non-randomized prospective observational study will be performed.

The recruited patients will undergo local injection of superficial enhanced fluid fat after a lower limb minor amputation. Laboratory analysis to evaluate the composition of the tissue and stromal cell components harvested from adipose tissue with SEFFICARE system by using digital droplets PCR. These data will serve for making associations between the clinical outcome and characteristics of the cell population administered to each patient.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFU) are one of the complications of diabetes mellitus resulting from multiple causes such as neuropathy, ischemia, and infection that contribute to morbidity and amputation. The prevalence of DFU has been estimated to be 3 to 5 times higher than the overall population. Minor amputations (digital or transmetatarsal) are the treatment of choice in case of irreversible DFU. However, many minor amputations do not heal and require re-amputation. Improvements of healing rate after adipose stem cells (ASCs) injection through micro-fragmented autologous adipose tissue of the amputation stump following minor DFU amputation were demonstrated. The use of ASCs obtained from the superficial enhanced fluid fat injection technique (SEFFICARE) to improve the healing process after DFUs minor amputation is the object of the present study.

STUDY DESIGN: Single-center non-randomized prospective observational cohort study.

TREATMENT: Local injection of superficial enhanced fluid fat after a lower limb minor amputation. Laboratory analysis to evaluate the composition of the tissue and stromal cell components harvested from adipose tissue with SEFFICARE system by using digital droplets PCR. These data will serve for making associations between the clinical outcome and characteristics of the cell population administered to each patient.

INCLUSION CRITERIA:

* type-1 and type-2 diabetes mellitus
* age >18-years
* both sexes
* chronic diabetic distal ulcers/gangrene (digital or forefoot) intended as W-grade 1 to 3 according to WifI classification;
* absence of active vascular issues or patients undergoing lower extremity revascularization to improve peripheral perfusion intended as I-grade 0 to 2 according to WIfi classification;
* absence of infection signs or presence of soft tissue infection intended as fI-grade 0 to 2 according to Wifi classification, without radiologic signs of bone infection (negative X-ray for osteolytic lesions); SAMPLE SIZE: The correct sample size was calculated considering as primary endpoint the proportion of the healing stump. The sample size was calculated with the Score Z test comparing one proportion based on literature results to a reference value. Using a significance level of 0.05, power of 0.8, setting the H0 proportion of 0.80 and the Ha of 0.6 respectively, the result was 36 subjects. An additional 10% of subjects was considered taking into account eventual drop-out during the study. The final sample size inflated to 40 patients.

ENDPOINTS: Primary endpoint: percentage of stump healing; Secondary endpoints:

* mean time for complete healing;
* evaluation of risk factors afflicting healing/failure;
* evaluation of reintervention (time elapsed since index operation, type, and indication);
* the prevalence of peripheral diabetic polyneuropathy at baseline;
* the percentage change in the pain score of NRS;
* health-related quality of life evaluation, intended as changing of the SF-36 score;
* collection of eventual adverse events related to the treatment procedure and eventual posthoc analysis.
* evaluation of the adipose harvested tissue composition and stromal cell components STATISTICAL ANALYSIS: The categorical endpoints, i.e., the difference in the healing rate will be assessed with the chi-square test or Fisher's exact test. The continuous variables will be calculated by Kaplan-Meier curves and log-rank test. A univariate and multivariate logistic regression analysis will be applied to identify influencing factors on the categorical endpoints. To test the influence of multiple variables on continuous data, one/two-way ANOVA will be performed with Bonferroni's post-test.

ELIGIBILITY:
Inclusion Criteria:

* type-1 and type-2 diabetes mellitus
* age >18-years
* both sexes
* chronic diabetic distal ulcers/gangrene (digital or forefoot) intended as W-grade 1 to 3 according to WifI classification;
* absence of active vascular issues or patients undergoing lower extremity revascularization to improve peripheral perfusion intended as I-grade 0 to 2 according to WIfi classification;
* absence of infection signs or presence of soft tissue infection intended as fI-grade 0 to 2 according to Wifi classification, without radiologic signs of bone infection (negative X-ray for osteolytic lesions);

Exclusion Criteria:

* extensive ulcers with deep involving proximal forefoot and/or deep, full-thickness heel ulcer, with calcaneal involvement (W-grade 3 according to WifI classification);
* active vascular issues [I-grade 3 according to Wifi classification];
* ulcers with signs of moderate and/or severe infection (osteomyelitis and/or sepsis) [fI-grade 3 according to WifI classification];
* severe comorbidities such as severe heart failure, liver failure, and/or psychiatric disorder;
* previous oncological treatments (past 5 years) or ongoing and/or neoplastic lesions;
* corticosteroid therapy;
* coagulopathy;
* infection of the harvesting site;
* local anesthetic allergy;
* immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Healing | 6 months
  Healing was defined as complete re-epithelialization of the stump after suture removal without signs of cutaneous suffering, inflammation, infection, local swelling as determined by one investigator.

SECONDARY OUTCOMES:
healing time change | 1, 2, 3, 4, 5, 6 months
  mean time for complete healing
risk factors afflicting healing/failure | 0 month
  evaluation of risk factors afflicting healing/failure
reintervention | 6 months
  time elapsed since index operation, type, and indication
diabetic peripheral neuropathy | 0 month
  the prevalence of DPN (probable) at baseline
health-related quality of life change | 1, 2, 3, 4, 5, 6 months
  health-related quality of life evaluation, intended as changing of the SF-36 score
adverse events related to the treatment procedure | 6 months
  collection of eventual adverse events related to the treatment procedure
amount of adipose stem cells used for grafting | 1 month
  amount of adipose stem cells used for grafting

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Silingardi, MD, Principal Investigator — University of Modena and Reggio Emilia; Manuela Simoni, MD, PhD, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- Ospedale Civile di Baggiovara (Modena), Azienda Ospedaliero-Universitaria di Modena, Università di Modena e Reggio Emilia, Modena, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvaro-Afonso FJ, Sanz-Corbalan I, Lazaro-Martinez JL, Kakagia D, Papanas N. Adipose-Derived Mesenchymal Stem Cells in the Treatment of Diabetic Foot Ulcers: A Review of Preclinical and Clinical Studies. Angiology. 2020 Oct;71(9):853-863. doi: 10.1177/0003319720939467. Epub 2020 Jul 29. PMID 32723090
- [Background] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- [Background] Zhang P, Lu J, Jing Y, Tang S, Zhu D, Bi Y. Global epidemiology of diabetic foot ulceration: a systematic review and meta-analysis dagger. Ann Med. 2017 Mar;49(2):106-116. doi: 10.1080/07853890.2016.1231932. Epub 2016 Nov 3. PMID 27585063
- [Background] Frykberg RG, Zgonis T, Armstrong DG, Driver VR, Giurini JM, Kravitz SR, Landsman AS, Lavery LA, Moore JC, Schuberth JM, Wukich DK, Andersen C, Vanore JV; American College of Foot and Ankle Surgeons. Diabetic foot disorders. A clinical practice guideline (2006 revision). J Foot Ankle Surg. 2006 Sep-Oct;45(5 Suppl):S1-66. doi: 10.1016/S1067-2516(07)60001-5. PMID 17280936
- [Background] Hingorani A, LaMuraglia GM, Henke P, Meissner MH, Loretz L, Zinszer KM, Driver VR, Frykberg R, Carman TL, Marston W, Mills JL Sr, Murad MH. The management of diabetic foot: A clinical practice guideline by the Society for Vascular Surgery in collaboration with the American Podiatric Medical Association and the Society for Vascular Medicine. J Vasc Surg. 2016 Feb;63(2 Suppl):3S-21S. doi: 10.1016/j.jvs.2015.10.003. PMID 26804367
- [Background] Prompers L, Huijberts M, Apelqvist J, Jude E, Piaggesi A, Bakker K, Edmonds M, Holstein P, Jirkovska A, Mauricio D, Ragnarson Tennvall G, Reike H, Spraul M, Uccioli L, Urbancic V, Van Acker K, van Baal J, van Merode F, Schaper N. High prevalence of ischaemia, infection and serious comorbidity in patients with diabetic foot disease in Europe. Baseline results from the Eurodiale study. Diabetologia. 2007 Jan;50(1):18-25. doi: 10.1007/s00125-006-0491-1. Epub 2006 Nov 9. PMID 17093942
- [Background] Prompers L, Schaper N, Apelqvist J, Edmonds M, Jude E, Mauricio D, Uccioli L, Urbancic V, Bakker K, Holstein P, Jirkovska A, Piaggesi A, Ragnarson-Tennvall G, Reike H, Spraul M, Van Acker K, Van Baal J, Van Merode F, Ferreira I, Huijberts M. Prediction of outcome in individuals with diabetic foot ulcers: focus on the differences between individuals with and without peripheral arterial disease. The EURODIALE Study. Diabetologia. 2008 May;51(5):747-55. doi: 10.1007/s00125-008-0940-0. Epub 2008 Feb 23. PMID 18297261
- [Background] Thorud JC, Jupiter DC, Lorenzana J, Nguyen TT, Shibuya N. Reoperation and Reamputation After Transmetatarsal Amputation: A Systematic Review and Meta-Analysis. J Foot Ankle Surg. 2016 Sep-Oct;55(5):1007-12. doi: 10.1053/j.jfas.2016.05.011. Epub 2016 Jul 27. PMID 27475711
- [Background] Uccioli L, Izzo V, Meloni M, Vainieri E, Ruotolo V, Giurato L. Non-healing foot ulcers in diabetic patients: general and local interfering conditions and management options with advanced wound dressings. J Wound Care. 2015 Apr;24(4 Suppl):35-42. doi: 10.12968/jowc.2015.24.Sup4b.35. PMID 25853647
- [Background] Vizoso FJ, Eiro N, Cid S, Schneider J, Perez-Fernandez R. Mesenchymal Stem Cell Secretome: Toward Cell-Free Therapeutic Strategies in Regenerative Medicine. Int J Mol Sci. 2017 Aug 25;18(9):1852. doi: 10.3390/ijms18091852. PMID 28841158
- [Background] Gimble JM, Guilak F, Bunnell BA. Clinical and preclinical translation of cell-based therapies using adipose tissue-derived cells. Stem Cell Res Ther. 2010 Jun 29;1(2):19. doi: 10.1186/scrt19. PMID 20587076
- [Background] Gadelkarim M, Abushouk AI, Ghanem E, Hamaad AM, Saad AM, Abdel-Daim MM. Adipose-derived stem cells: Effectiveness and advances in delivery in diabetic wound healing. Biomed Pharmacother. 2018 Nov;107:625-633. doi: 10.1016/j.biopha.2018.08.013. Epub 2018 Aug 14. PMID 30118878
- [Background] Zuk PA, Zhu M, Ashjian P, De Ugarte DA, Huang JI, Mizuno H, Alfonso ZC, Fraser JK, Benhaim P, Hedrick MH. Human adipose tissue is a source of multipotent stem cells. Mol Biol Cell. 2002 Dec;13(12):4279-95. doi: 10.1091/mbc.e02-02-0105. PMID 12475952
- [Background] Caruana G, Bertozzi N, Boschi E, Pio Grieco M, Grignaffini E, Raposio E. Role of adipose-derived stem cells in chronic cutaneous wound healing. Ann Ital Chir. 2015 Jan-Feb;86(1):1-4. PMID 25818696
- [Background] Salgado AJ, Reis RL, Sousa NJ, Gimble JM. Adipose tissue derived stem cells secretome: soluble factors and their roles in regenerative medicine. Curr Stem Cell Res Ther. 2010 Jun;5(2):103-10. doi: 10.2174/157488810791268564. PMID 19941460
- [Background] Arcidiacono JA, Blair JW, Benton KA. US Food and Drug Administration international collaborations for cellular therapy product regulation. Stem Cell Res Ther. 2012 Sep 28;3(5):38. doi: 10.1186/scrt129. PMID 23021082
- [Background] Gutowski KA; ASPS Fat Graft Task Force. Current applications and safety of autologous fat grafts: a report of the ASPS fat graft task force. Plast Reconstr Surg. 2009 Jul;124(1):272-280. doi: 10.1097/PRS.0b013e3181a09506. PMID 19346997
- [Background] Yoshimura K, Shigeura T, Matsumoto D, Sato T, Takaki Y, Aiba-Kojima E, Sato K, Inoue K, Nagase T, Koshima I, Gonda K. Characterization of freshly isolated and cultured cells derived from the fatty and fluid portions of liposuction aspirates. J Cell Physiol. 2006 Jul;208(1):64-76. doi: 10.1002/jcp.20636. PMID 16557516
- [Background] Lonardi R, Leone N, Gennai S, Trevisi Borsari G, Covic T, Silingardi R. Autologous micro-fragmented adipose tissue for the treatment of diabetic foot minor amputations: a randomized controlled single-center clinical trial (MiFrAADiF). Stem Cell Res Ther. 2019 Jul 29;10(1):223. doi: 10.1186/s13287-019-1328-4. PMID 31358046
- [Background] Bernardini FP, Gennai A, Izzo L, Zambelli A, Repaci E, Baldelli I, Fraternali-Orcioni G, Hartstein ME, Santi PL, Quarto R. Superficial Enhanced Fluid Fat Injection (SEFFI) to Correct Volume Defects and Skin Aging of the Face and Periocular Region. Aesthet Surg J. 2015 Jul;35(5):504-15. doi: 10.1093/asj/sjv001. Epub 2015 Apr 24. PMID 25911629
- [Background] Bernardini FP, Gennai A. Fluid Fat Injection for Volume Restoration and Skin Regeneration of the Periocular Aesthetic Unit. JAMA Facial Plast Surg. 2016 Jan-Feb;18(1):68-70. doi: 10.1001/jamafacial.2015.1146. No abstract available. PMID 26587895
- [Background] Gennai A, Zambelli A, Repaci E, Quarto R, Baldelli I, Fraternali G, Bernardini FP. Skin Rejuvenation and Volume Enhancement with the Micro Superficial Enhanced Fluid Fat Injection (M-SEFFI) for Skin Aging of the Periocular and Perioral Regions. Aesthet Surg J. 2017 Jan;37(1):14-23. doi: 10.1093/asj/sjw084. Epub 2016 May 30. PMID 27241362
- [Background] Rossi M, Roda B, Zia S, Vigliotta I, Zannini C, Alviano F, Bonsi L, Zattoni A, Reschiglian P, Gennai A. Characterization of the Tissue and Stromal Cell Components of Micro-Superficial Enhanced Fluid Fat Injection (Micro-SEFFI) for Facial Aging Treatment. Aesthet Surg J. 2020 May 16;40(6):679-690. doi: 10.1093/asj/sjy142. PMID 29905790
- [Background] Lazarus GS, Cooper DM, Knighton DR, Margolis DJ, Pecoraro RE, Rodeheaver G, Robson MC. Definitions and guidelines for assessment of wounds and evaluation of healing. Arch Dermatol. 1994 Apr;130(4):489-93. PMID 8166487
- [Background] Sheehan P, Jones P, Giurini JM, Caselli A, Veves A. Percent change in wound area of diabetic foot ulcers over a 4-week period is a robust predictor of complete healing in a 12-week prospective trial. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):239S-244S. doi: 10.1097/01.prs.0000222891.74489.33. PMID 16799391
- [Background] Cardenas-Camarena L. Lipoaspiration and its complications: a safe operation. Plast Reconstr Surg. 2003 Oct;112(5):1435-41; discussion 1442-3. doi: 10.1097/01.PRS.0000081469.07342.F2. PMID 14504529
- [Background] Mills JL Sr, Conte MS, Armstrong DG, Pomposelli FB, Schanzer A, Sidawy AN, Andros G; Society for Vascular Surgery Lower Extremity Guidelines Committee. The Society for Vascular Surgery Lower Extremity Threatened Limb Classification System: risk stratification based on wound, ischemia, and foot infection (WIfI). J Vasc Surg. 2014 Jan;59(1):220-34.e1-2. doi: 10.1016/j.jvs.2013.08.003. Epub 2013 Oct 12. PMID 24126108
- [Background] Monteiro-Soares M, Russell D, Boyko EJ, Jeffcoate W, Mills JL, Morbach S, Game F; International Working Group on the Diabetic Foot (IWGDF). Guidelines on the classification of diabetic foot ulcers (IWGDF 2019). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3273. doi: 10.1002/dmrr.3273. PMID 32176445
- [Background] Feldman EL, Stevens MJ, Thomas PK, Brown MB, Canal N, Greene DA. A practical two-step quantitative clinical and electrophysiological assessment for the diagnosis and staging of diabetic neuropathy. Diabetes Care. 1994 Nov;17(11):1281-9. doi: 10.2337/diacare.17.11.1281. PMID 7821168
- [Background] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709
- [Background] Schaper NC, Van Netten JJ, Apelqvist J, Lipsky BA, Bakker K; International Working Group on the Diabetic Foot (IWGDF). Prevention and management of foot problems in diabetes: A Summary Guidance for Daily Practice 2015, based on the IWGDF guidance documents. Diabetes Res Clin Pract. 2017 Feb;124:84-92. doi: 10.1016/j.diabres.2016.12.007. Epub 2016 Dec 18. PMID 28119194
- [Background] Danielsson M, Halvardson J, Davies H, Torabi Moghadam B, Mattisson J, Rychlicka-Buniowska E, Jaszczynski J, Heintz J, Lannfelt L, Giedraitis V, Ingelsson M, Dumanski JP, Forsberg LA. Longitudinal changes in the frequency of mosaic chromosome Y loss in peripheral blood cells of aging men varies profoundly between individuals. Eur J Hum Genet. 2020 Mar;28(3):349-357. doi: 10.1038/s41431-019-0533-z. Epub 2019 Oct 25. PMID 31654039
- [Background] Casarini L, Lazzaretti C, Paradiso E, Limoncella S, Riccetti L, Sperduti S, Melli B, Marcozzi S, Anzivino C, Sayers NS, Czapinski J, Brigante G, Poti F, La Marca A, De Pascali F, Reiter E, Falbo A, Daolio J, Villani MT, Lispi M, Orlando G, Klinger FG, Fanelli F, Rivero-Muller A, Hanyaloglu AC, Simoni M. Membrane Estrogen Receptor (GPER) and Follicle-Stimulating Hormone Receptor (FSHR) Heteromeric Complexes Promote Human Ovarian Follicle Survival. iScience. 2020 Nov 18;23(12):101812. doi: 10.1016/j.isci.2020.101812. eCollection 2020 Dec 18. PMID 33299978
- [Background] Bourin P, Bunnell BA, Casteilla L, Dominici M, Katz AJ, March KL, Redl H, Rubin JP, Yoshimura K, Gimble JM. Stromal cells from the adipose tissue-derived stromal vascular fraction and culture expanded adipose tissue-derived stromal/stem cells: a joint statement of the International Federation for Adipose Therapeutics and Science (IFATS) and the International Society for Cellular Therapy (ISCT). Cytotherapy. 2013 Jun;15(6):641-8. doi: 10.1016/j.jcyt.2013.02.006. Epub 2013 Apr 6. PMID 23570660
- [Background] Dominici M, Le Blanc K, Mueller I, Slaper-Cortenbach I, Marini F, Krause D, Deans R, Keating A, Prockop Dj, Horwitz E. Minimal criteria for defining multipotent mesenchymal stromal cells. The International Society for Cellular Therapy position statement. Cytotherapy. 2006;8(4):315-7. doi: 10.1080/14653240600855905. PMID 16923606
- [Background] Fink T, Lund P, Pilgaard L, Rasmussen JG, Duroux M, Zachar V. Instability of standard PCR reference genes in adipose-derived stem cells during propagation, differentiation and hypoxic exposure. BMC Mol Biol. 2008 Oct 31;9:98. doi: 10.1186/1471-2199-9-98. PMID 18976469